CLINICAL TRIAL: NCT01961102
Title: Pilot-study of OSCAR ENDO One Stop Assessment of Risk for Endometrial Hyperplasia and Cancer
Brief Title: OSCAR ENDO One Stop Assessment of Risk for Endometrial Hyperplasia and Cancer
Status: Completed | Type: Observational
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Other Study IDs: BHS-Gyn1
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2015-12

CONDITIONS: Endometrial Cancer; Atypical Hyperplasia
Keywords: postmenopausal bleeding; postmenopausal hyperplasia; endometrial cancer; atypical hyperplasia; curettage; intraoperative rapid section
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Hysteroscopy; Curettage

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: hysteroscopy/curettage in case of suspicious aspect will be done a rapid section
  Other Names: OSCAR Endo Study

SUMMARY:
It is to be achieved that in postmenopausal women through the combination of Hysteroscopy and intraoperative rapid section a positive predictive value (PPV) regarding the objective illness like endometrial cancer or adenomatous hyperplasia of 100% so as a negative predictive value (NPV) of 99%.

DETAILED DESCRIPTION:
If a patient fulfills the inclusion criteria, the surgeon decides intraoperatively due to the aspect in the hysteroscopy if it is a clearly benign result or if it looks suspicious or malign.

In case of a hysteroscopical benign result the patient will be informed about the result after the operation.

In case of a hysteroscopal suspicious or malignant aspect, the curettement will be sent for a rapid section. If the hysteroscopic result confirms the hysteroscopic suspicion the patient will be informed after the operation and the further treatment can be planned right away.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status (more than 1 year of last menopausal bleeding)
* Postmenopausal vaginal bleeding
* Asymptomatic postmenopausal endometrial hyperplasia
* Understanding of the german language
* Signature and consent of the patient

Exclusion Criteria:

* Not able to understand and participate in the study
* Premenopausal status
* no informed consent

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
A negative predictive value of 99 % | Intraoperative
  To get in combination of hysteroscopy and rapid section of the endometrial curettement a negative predictive value of 99% as well as a positive predictive value of 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynaecology, Barmherzige Schwestern, Linz, Austria

REFERENCES:
- [Derived] Hefler-Frischmuth K, Hirtl-Goergl E, Unterrichter V, Lafleur J, Brunnmayr-Petkin G, Moinfar F, Hefler L. One-stop clinical assessment of risk for endometrial hyperplasia (OSCAR-Endo): a fast-track protocol for evaluating endometrial pathologies. Arch Gynecol Obstet. 2017 Apr;295(4):959-964. doi: 10.1007/s00404-017-4326-8. Epub 2017 Mar 6. PMID 28265757